CLINICAL TRIAL: NCT00524420
Title: Transcranial Magnetic Stimulation (TMS) in the Treatment of Chronic Widespread Pain (CWP)
Brief Title: Transcranial Magnetic Stimulation for Treating Women With Chronic Widespread Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, David Avery, Study Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 32656-D; R21AR053963 (NIH); 1R21AR053963-01 (NIH); 06-2407-D 01 (Other: UW Human Subjects Division ID)
Record Dates: First submitted 2007-08-30; First posted 2007-09-03 (Estimated); Results first posted 2013-05-23 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-04

CONDITIONS: Fibromyalgia; Chronic Pain; Depression
Keywords: Pain; Fatigue; Chronic Fatigue Syndrome; Chronic Fatigue-Fibromyalgia Syndrome; Depression; Major Depressive Disorder
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Depression; Pain; Fatigue; Fatigue Syndrome, Chronic; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active rTMS (Experimental): Active rTMS involves administration of real rTMS to the patient.
  Interventions: Device: rTMS
- Sham rTMS (Sham Comparator): Sham rTMS is a placebo or inactive form of rTMS for study control and comparison purposes.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: rTMS — 10 Hz, 4-second trains, 26-second intertrain interval, 75 trains/session, 15 sessions at 120% motor threshold rTMS to left dorsolateral prefrontal cortex
  Other Names: Neuronetics 2100 CRS rTMS System
  Arms: Active rTMS
Device: Sham rTMS — 10 Hz, 4-second trains, 26-second intertrain interval, 75 trains/session, 15 sessions of sham rTMS
  Other Names: Neuronetics 2100 rTMS and James Long Integrated Sham System
  Arms: Sham rTMS

SUMMARY:
While acute pain after surgery or trauma comes on suddenly and lasts for a limited amount of time, chronic pain persists and can continue for months and even years. Repetitive transcranial magnetic stimulation (rTMS) uses a magnetic field to deliver a current to the brain and can affect brain activity. The purpose of this study is to determine the effectiveness of rTMS treatment in reducing chronic widespread pain in women.

DETAILED DESCRIPTION:
Chronic widespread pain is characterized by musculoskeletal pain that lasts for at least 3 months, pain above and below the waist, pain on both the right and left sides, and pain in the head, neck, spine, or back. In addition to fatigue, chronic widespread pain is a hallmark feature of fibromyalgia. Significant physical and emotional effects usually accompany chronic widespread pain and fibromyalgia, making the development of effective treatments a priority. rTMS involves a neurophysiologic technique that directs a current into the brain by using a magnetic field to pass the scalp and skull safely and painlessly. Stimuli are applied to the same brain area several times per second during several consecutive seconds. rTMS has been found to be effective for treating certain types of chronic pain. The purpose of this study is to determine the effectiveness of rTMS treatment in reducing bodily pain associated with chronic widespread pain and/or fibromyalgia in women.

Participants in this study will undergo a diagnostic interview, physical and neurological exam, electrocardiogram, magnetic resonance imaging, and blood and urine collection for screening purposes. Eligible participants will then be randomly assigned to receive either rTMS treatment or sham rTMS treatment. One-hour daily treatment sessions will occur over 15 days. After every five treatment sessions, participants will be interviewed about their pain and depression symptoms, and they will fill out questionnaires about pain, depression, fatigue, sleep, and exercise. Participants will also undergo pain threshold and tolerance testing of their right thumb. On a daily basis, participants will rate their level of pain using a 0 to 20 scale. Follow-up evaluations will occur 1, 4, and 12 weeks after treatment and will include a repeat interview and testing. After the follow-up evaluations, any participants who did not respond to the sham treatment will be offered a series of 15 real rTMS treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic widespread pain as defined by the 1990 American College of Rheumatology guidelines: chronic musculoskeletal pain for at least 3 months; pain above and below the waist; pain on both right and left sides; pain at one axial site (e.g., head, neck, spine, or back)
* Willing to remain on a stable medical regimen during the entire 6-week course of Phase 1 treatment and 8 weeks prior to rTMS treatment
* Willing to undergo random assignment and able to attend treatment sessions
* Willing to remain on a stable psychotherapy regimen if currently receiving psychotherapy that has been ongoing for at least 3 months prior to study entry

Exclusion Criteria:

* Unable to maintain treatment as usual at stable doses for any medical or psychiatric conditions for 8 weeks prior to and during the study
* Another medical condition associated with significant pain (e.g., diabetic neuropathy, systemic lupus erythematosus, Rheumatoid arthritis, severe degenerative joint disease)
* Any condition that might increase the risk of seizures from TMS
* History of a seizure disorder or family history of a seizure disorder
* Previous use of TMS
* Involvement in litigation or disability that is related to fibromyalgia, chronic widespread pain, or depression
* Current use of proconvulsant medications (e.g., bupropion)
* Metal in the body that would prevent magnetic resonance imaging (MRI) or TMS (e.g., aneurysm clips, pacemakers, neurostimulators)
* History of head injury associated with loss of consciousness for more than 15 minutes, brain surgery, or lithium toxicity
* History of bipolar disorder, schizophrenia, obsessive compulsive disorder, panic disorder, or post-traumatic stress disorder
* Current substance abuse or dependence
* Active suicidal intent or plan
* Severe claustrophobia that would prevent MRI
* Major depression with psychotic features or a current major depressive episode lasting longer than 5 years
* Pregnant

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Avery, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Avery DH, Holtzheimer PE 3rd, Fawaz W, Russo J, Neumaier J, Dunner DL, Haynor DR, Claypoole KH, Wajdik C, Roy-Byrne P. Transcranial magnetic stimulation reduces pain in patients with major depression: a sham-controlled study. J Nerv Ment Dis. 2007 May;195(5):378-81. doi: 10.1097/NMD.0b013e31802f58d1. PMID 17502802
- See also: Click here for the Neuronetics, Inc. Homepage — http://www.neuronetics.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between January 2008 and November 2010. Subjects were recruited from advertisements, referrals, and from a University of Washington clinic that specializes in Fibromyalgia.
Pre-assignment Details: 493 subjects were screened over the phone. 31 subjects came into the clinic for an initial screening visit. Subjects were allowed to maintain stable doses of medication and psychotherapy. 12 of the screened subjects did not meet criteria for randomization. The remaining 19 were randomized, and 18 completed the study.
Groups:
- Active rTMS: rTMS : 10 Hz, 4-second trains, 26-second intertrain interval, 75 trains/session, 15 sessions at 120% motor threshold rTMS to left dorsolateral prefrontal cortex
- Sham rTMS: Sham rTMS : 10 Hz, 4-second trains, 26-second intertrain interval, 75 trains/session, 15 sessions of sham rTMS
Period: Overall Study
Arm/Group | Active rTMS | Sham rTMS
Started | 8 (One was incorrectly randomized;she did not have a BIRS of >7. Was excluded from efficacy analysis.) | 11
Completed | 7 (1 dropped out after treatment 10 because of poor response and was included in the efficacy analyses.) | 11
Not Completed | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS | Sham rTMS | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 11 | 19
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 54.86 (7.65) | 52.09 (10.02) | 53.17 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Gracely Box Intensity Rating Scale
Description: The BIRS is reliable, valid, and sensitive measure that has been used in a number of studies of analgesics and studies of changes of pain intensity over time and was selected as the primary outcome variable. Each scale is a 20 point scale that has clear anchor points. Patients will be classified as responders if they have a 4 point drop or more on the BIRS. In order to be randomized, subjects were to have had a BIRS score of at least 8. Lower scores indicate less pain and higher scores indicate more pain. This measure was administered once a week at Baseline, at the end of weeks 1, 2, and 3 of TMS treatment, and 1 week post-TMS treatment.
Time Frame: Measured weekly
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham rTMS | Active rTMS
Number analyzed (Participants) | 11 | 7
units on a scale
  Baseline | 13.18 (2.79) | 14.43 (2.23)
  TMS Treatment Week 1 | 10.64 (3.41) | 13.00 (3.46)
  TMS Treatment Week 2 | 10.27 (3.80) | 11.29 (4.75)
  TMS Treatment Week 3 | 8.45 (5.11) | 10.58 (6.07)
  1 Week Post TMS | 8.60 (5.56) | 10.50 (5.96)

2. Secondary Outcome: Gracely Box Unpleasantness Scale
Description: The BURS is reliable, valid, and sensitive measure that has been used in a number of studies of analgesics and studies of changes of pain unpleasantness over time. Each scale is a 20 point scale that has clear anchor points. Pain unpleasantness is different from pain intensity in that it assesses the affective and not the somatic aspect of the pain. Lower scores indicate less unpleasantness of pain and higher scores indicate more unpleasantness of pain. This measure was administered at Baseline, after weeks 1, 2, and 3 of TMS treatment, and 1 week post-TMS.
Time Frame: Measured weekly
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham rTMS | Active rTMS
Number analyzed (Participants) | 11 | 7
units on a scale
  Baseline | 9.91 (2.77) | 12.57 (1.72)
  TMS Treatment Week 1 | 8.73 (3.32) | 11.86 (4.38)
  TMS Treatment Week 2 | 9.00 (3.85) | 10.43 (4.61)
  TMS Treatment Week 3 | 7.73 (4.13) | 9.50 (6.50)
  1 Week Post TMS | 7.60 (4.84) | 9.83 (6.05)

3. Secondary Outcome: Hamilton Depression Rating Scale
Description: The research coordinator administered the Hamilton Depression Rating Scale-17 item to assess the level of depression on a weekly basis at baseline, weeks 1, 2, 3 of TMS treatment and 1 week post-TMS treatment. Higher scores indicate a higher level of depression. Scores range from 0-50 and scores greater than 20 generally indicate moderate depression. Scores between 0-7 are considered normal.
Time Frame: Measured weekly
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham rTMS | Active rTMS
Number analyzed (Participants) | 11 | 7
units on a scale
  Baseline | 14.64 (6.34) | 14.71 (6.55)
  TMS Treatment Week 1 | 11.18 (6.60) | 15.43 (5.38)
  TMS Treatment Week 2 | 9.09 (5.13) | 11.86 (5.96)
  TMS Treatment Week 3 | 8.36 (5.01) | 10.83 (5.78)
  1 Week Post TMS | 7.45 (4.30) | 8.67 (6.25)

4. Secondary Outcome: Adverse Events
Description: Adverse events (AEs) were collected by open report of emergent symptoms or illness during the study. This form is filled out during baseline, daily before each TMS session by the trained physician administering the TMS, and at each follow-up visit.
Time Frame: Measured daily
Measure: Number; unit: number of adverse events
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 8 | 11
number of adverse events | 36 | 35

ADVERSE EVENTS:
Arm/Group | Active rTMS | Sham rTMS
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 5/8 | 5/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active rTMS (N=8) | Sham rTMS (N=11)
pain at the site of stimulation (Injury, poisoning and procedural complications) | 4 | 3
increased muscle aches (Musculoskeletal and connective tissue disorders) | 2 | 1
increased fatigue (Musculoskeletal and connective tissue disorders) | 1 | 1
headache (Nervous system disorders) | 5 | 5
insomnia (Nervous system disorders) | 2 | 1
tingling sensation in scalp during stimulation (Injury, poisoning and procedural complications) | 0 | 1
dizziness (Nervous system disorders) | 1 | 1
confusion (Nervous system disorders) | 0 | 1
tiredness after session (Musculoskeletal and connective tissue disorders) | 0 | 1
shakiness (Nervous system disorders) | 1 | 0
anxiety (Psychiatric disorders) | 1 | 0
lightheadedness after session (Injury, poisoning and procedural complications) | 1 | 0
poor concentration (Psychiatric disorders) | 1 | 0
"fuzzy-headed" after TMS (Psychiatric disorders) | 1 | 0
migraine (Nervous system disorders) | 1 | 0
pain in teeth during stimulation (Injury, poisoning and procedural complications) | 0 | 1
drowsiness (Nervous system disorders) | 0 | 1
feeling more "distant, detached" (Psychiatric disorders) | 0 | 1
flat affect (Psychiatric disorders) | 0 | 1
twitching of eye (Injury, poisoning and procedural complications) | 0 | 1
pain in jaw (Injury, poisoning and procedural complications) | 0 | 1
sore throat (Infections and infestations) | 1 | 1
coryza (Infections and infestations) | 1 | 0
cough (Infections and infestations) | 1 | 1
sinus headache (Infections and infestations) | 1 | 0
flu (Infections and infestations) | 2 | 0
viral infection (Infections and infestations) | 1 | 0
tinnitus (Ear and labyrinth disorders) | 1 | 1
sinus infection (Infections and infestations) | 0 | 1
dry mouth (General disorders) | 0 | 1
sinus congestion (Infections and infestations) | 0 | 1
sinus drainage (Infections and infestations) | 0 | 1
nausea (Gastrointestinal disorders) | 2 | 1
abdominal pain (Gastrointestinal disorders) | 2 | 1
diarrhea (Gastrointestinal disorders) | 1 | 0
sebaceous cyst on thigh (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TMJ pain (Injury, poisoning and procedural complications) | 1 | 0
heart palpitations (Cardiac disorders) | 0 | 2
dry eyes (Eye disorders) | 0 | 1
pain in thumb (Musculoskeletal and connective tissue disorders) | 0 | 1
pain in shoulder (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No